CLINICAL TRIAL: NCT06652997
Title: SPH3348 Tablets in a Single-center, Randomized, Open-label, Single-dose, Two-period, Two-sequence Crossover Design Food Effect Study in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Collaborators: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Principal Investigator, Yu Qin, Principal Investigator, West China Second University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SPH3348-102
Record Dates: First submitted 2024-10-16; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Antitumor Drug; Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Randomized, Open-label, Single-dose, Two-period, Two-sequence Crossover Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single oral administration of SPH3348 tablets under fasting condition (Active Comparator): Single oral administration of SPH3348 tablets（480 mg） under fasting condition
  Interventions: Drug: SPH3348
- Single oral administration of SPH3348 tablets under fed condition (Active Comparator): Single oral administration of SPH3348 tablets（480 mg） under fed condition
  Interventions: Drug: SPH3348

INTERVENTIONS:
Drug: SPH3348 — Single oral administration of SPH3348 tablets（480mg） under fasting and fed conditions

SUMMARY:
The goal of this clinical trial is to evaluate the pharmacokinetic (PK) characteristics of single oral doses of SPH3348 tablets in healthy subjects under fasting and fed conditions, as well as the impact of food on PK.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for this trial, participants must meet all the following inclusion criteria:

  1. Fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial, and sign an informed consent form, being able to complete all trial processes as required by the protocol;
  2. Be healthy adult males or females aged 18 to 45 years, inclusive of the boundary values;
  3. Have a body mass index (BMI) of 18 to 26 kg/m^2, inclusive of the boundary values, with a minimum weight of 50 kg for males and 45 kg for females;
  4. Participants with potential for fertility must use at least one medically recognized contraceptive method during the study treatment period and for one year after the end of the study treatment (contraceptive methods and requirements are detailed in Appendix 1); females must undergo a pregnancy test during the screening period or at admission, with a result that must be negative; and must not be breastfeeding.

Exclusion Criteria:

* Participants who meet any of the following exclusion criteria will be excluded:

  1. Have a history of clinically significant diseases in the heart, liver, kidney, respiratory, hematopoietic, nervous, urinary reproductive systems, or mental diseases, severe infections, severe trauma, or major surgical procedures within 3 months before administration, or plan to undergo surgical procedures during the study;
  2. Have a history of suspected allergy to the study drug or any component of the study drug (including drug allergies and food allergies, etc.);
  3. Have a history of diseases or have received treatments that affect the absorption, distribution, metabolism, and excretion of drugs in the body, as determined by the investigator, such as gastrectomy, gastrointestinal anastomosis, laparoscopic Roux-en-Y gastric bypass surgery, etc.;
  4. Have difficulty with venous blood collection or have a history of fainting from needles or blood or physical conditions that cannot withstand intensive blood collection;
  5. Have an average daily smoking consumption of more than 5 cigarettes in the 3 months before screening or are unable to give up the use of tobacco products during the entire trial period;
  6. Have a history of drug use, a history of drug abuse (such as THC, morphine, ketamine, methamphetamine, MDMA) within 6 months before screening, or have a positive urine drug screen;
  7. Consume more than 14 units of alcohol per week in the 6 months before screening (1 standard unit = 14 g of alcohol = 360 mL of beer or 45 mL of liquor with 40% alcohol or 150 mL of wine) or are unable to abstain from alcohol during the trial period, or have an abnormal alcohol breath test (acceptable range: 0~3 mg/100 mL);
  8. Have used any prescription drugs, over-the-counter drugs, Chinese herbal medicine, or health products within 4 weeks before the start of the trial;
  9. Be vegetarians, have dietary restrictions that cannot comply with a uniform diet, or have difficulty swallowing;
  10. Have consumed foods that affect liver enzymes (such as grapefruit and grapefruit-containing products) or any foods rich in xanthine substances (such as coffee, tea, chocolate, cocoa, milk tea, etc.) within 48 hours before taking medication, or have engaged in vigorous exercise;
  11. Test positive for Hepatitis B surface antigen (HBsAg), Hepatitis C virus antibody (HCV-Ab), Human Immunodeficiency Virus antibody (HIV-Ab), or syphilis antibody;
  12. Have abnormal results in vital sign assessment, physical examination, laboratory tests, 12-lead ECG, and chest PA X-ray that are clinically significant;
  13. Have a corrected QT interval (QTcB) obtained from a 12-lead ECG at rest of >450 ms in males and >470 ms in females at screening, or have other abnormalities deemed clinically significant by the investigator;
  14. Have participated in other drug or medical device clinical trials within 3 months before screening;
  15. Have received or plan to receive live (attenuated) vaccines during the trial process or within one month after administration;
  16. Have donated blood or lost a total of ≥200 mL of blood within 1 month before screening, or have donated blood or lost ≥400 mL within 3 months before administration; have received blood transfusions or blood products;
  17. Are deemed ineligible for enrollment by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Cmax | Cmax occurs within 1.5 to 4 hours after dosing
  Peak Concentration
Tmax | From administration to reaching maximum plasma concentration, typically around 3 hours
  "Time to Reach Maximum Concentration
AUC0-t | AUC0-t is measured from time 0 to 32 hours post-dose

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 17 days

CONTACTS AND LOCATIONS:
Overall Officials: yu, Principal Investigator — National Drug Clinical Trial Institution of West China Second Hospital
Locations (1):
- West China Second University Hospital, Chengdu, China